CLINICAL TRIAL: NCT05555121
Title: Rescue Progesterone Supplementation in Patients With Low Progesterone on the Day of Embryo Transfer for Artificial Endometrial Preparation Cycles: a Non-inferiority Study
Brief Title: Rescue Progesterone Supplementation During Frozen Embryo Transfer
Acronym: P4R
Status: Suspended | Phase: Phase 2 | Type: Interventional
Why Stopped: Study medication temporarly not available in Canada.
Sponsor: Clinique Ovo (Industry)
Collaborators: Ferring Pharmaceuticals (Industry)
Responsible Party: Sponsor
Allocation: Non-Randomized | Model: Parallel | Masking: None | Purpose: Treatment
Other Study IDs: IIS-1032
Record Dates: First submitted 2022-09-16; First posted 2022-09-26 (Actual); Last update posted 2025-12-09 (Actual); Status verified 2025-12

CONDITIONS: Fertility Issues; Embryo Implantation; Frozen Embryo Transfer
Keywords: Embryo; Frozen embryo transfer; Progesterone; Embryo implantation
MeSH Terms: conditions — Infertility | interventions — Progesterone

STUDY DESIGN:
Intervention Model Description: Single centre, prospective, open label study
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No | US Export: No

ARMS (2):
- Endometrin 100 mg three times per day (TID) (Active Comparator): Women with progesterone levels ≥ 8.8 ng/ml during frozen embryo transfer cycle will take Endometrin 100 mg TID until 10th week of pregnancy
  Interventions: Drug: Progesterone Effervescent Vaginal Tablet
- Endometrin 200 mg three times per day (TID) (Active Comparator): Women with progesterone levels < 8.8 ng/ml during frozen embryo transfer cycle will take Endometrin 200 mg TID until 10th week of pregnancy
  Interventions: Drug: Progesterone Effervescent Vaginal Tablet

INTERVENTIONS:
Drug: Progesterone Effervescent Vaginal Tablet — On the day of Frozen Embryo Transfer (FET), women will have a blood test to determine progesterone levels. Depending on the result of progesterone level, the participant will be assigned to either the Endometrin 100 mg TID dose or the Endometrin 200 mg TID dose
  Other Names: Endometrin

SUMMARY:
Endometrin is a progesterone supplement prescribed during in vitro fertilization (IVF) for preparation for embryo transfer. The usual dose of Endometrin is 100 mg two to three times per day in the form of an effervescent tablet to be inserted vaginally.

The purpose of this research project is to evaluate the dose response of the Endometrin when determined based on the blood level of progesterone on the day of the FET. According to the literature, a predefined level of progesterone in the blood should be reached in order to have favorable conditions for pregnancy. The hypothesis being that a woman with low progesterone levels would benefit from a dose of Endometrin of 600 mg (200 mg 3x/day) to decrease the risk of miscarriage and improve the chances of pregnancy. Women with adequate progesterone levels according to the literature, would continue with the standard dose of progesterone prescribed at clinique ovo which is 300 mg (100 mg 3x/day).

PIBF (Progesterone Induced Blocking Factor) levels, a protein found in the blood that could also predict pregnancy outcomes in women using IVF will also be looked at.

ELIGIBILITY:
Inclusion Criteria:

* Women 18-42 years of age
* Normal uterine cavity (according to treating physician)
* FET substituted cycle prescribed
* First or second cycle of FET
* Adequate endometrial pattern (triple layer) and thickness (>7 mm) after adequate standard endometrial preparation in artificial cycle

Exclusion Criteria:

* Any uterine abnormalities confirmed by treating physician making participant unable to proceed with FET
* Patients with personalized FET according to the endometrial receptivity assay tests
* Previous allergic reactions to progesterone or any of the ingredients of Endometrin
* Severe hepatic dysfunction or disease
* Known or suspected breast cancer or genital tract cancer
* Known active arterial or venous thromboembolism or severe thrombophlebitis or cerebro-vascular disease, or a history of these events
* Diagnosed porphyria
* Undiagnosed abnormal vaginal bleeding
* Known missed abortion or ectopic pregnancy
* Recurrent pregnancy loss excluding biochemical pregnancies
* Hypersensitivity to Acetylsalicylic acid (ASA), salicylates, non-steroidal anti-inflammatory drugs (NSAIDs), analgesics, antipyretics or other ingredients in the product or component of the container
* Acute gastrointestinal ulcer, history of gastrointestinal ulcers and hemorrhagic diathesis
* Active or severe renal disease, or congestive heart failure
* History of asthma induced by salicylates or other NSAIDs
* Use of methotrexate at doses of 15mg/week or more
* Glucose-6-phosphate dehydrogenase (G6PD) deficiency

Ages: 18 Years to 42 Years | Sex: Female | Healthy Volunteers: No
Age Groups: Adult
Gender Based: Yes
Enrollment: 150 (Estimated)
Dates: Start 2022-12-01 (Actual); Primary Completion 2028-04-30 (Estimated); Study Completion 2028-06-30 (Estimated)

PRIMARY OUTCOMES:
Evaluate the ongoing pregnancy rate | 6 to 8 weeks after Frozen Embryo Transfer
  Viability ultrasound

SECONDARY OUTCOMES:
Evaluate the miscarriage rate | 6 to 8 weeks after Frozen Embryo Transfer
  Viability ultrasound
Evaluate progesterone levels | Before embryo transfer and 10 days after embryo transfer
  Progesterone levels will be tested at two different times
Evaluate the rate of biochemical pregnancy | 10 days after frozen embryo transfer
  Serum pregnancy test to measure Beta Human Chorionic Gonadotropin (BhCG) levels

OTHER OUTCOMES:
Blood test to evaluate the prevalence of PIBF | Before embryo transfer and 10 days after embryo transfer
  Progesterone Inducing Blocking Factor (PIBF) has been found to to have an important part in creating a welcoming environment for the embryo

CONTACTS AND LOCATIONS:
Overall Officials: Wael Jamal, MD, Principal Investigator — Clinique Ovo
Locations (1):
- Clinique Ovo, Montreal, Quebec, Canada

IPD SHARING:
Plan to Share IPD: No